CLINICAL TRIAL: NCT07372274
Title: The Effects of Glenohumeral Internal Rotation Deficit on Posterior Shoulder Endurance and Upper Extremity Stability in Adolescent Male Volleyball Players
Brief Title: Effect of Glenohumeral Internal Rotation Deficit on Shoulder Endurance and Stability in Adolescent Male Volleyball Players
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Seda Uluşahin, Principal Investigator, PT PhD, Saglik Bilimleri Universitesi
Other Study IDs: 2024-534
Record Dates: First submitted 2026-01-13; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Glenohumeral Internal Rotation Deficit (GIRD)
Keywords: Glenohumeral internal rotation deficit; adolescent athletes; volleyball players

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Glenohumeral internal rotation deficit (GIRD) Group: GIRD Present (≥10° internal rotation deficit)
  Interventions: Other: Glenohumeral Rotation ROM, Shoulder Endurance, and Upper Extremity Stability Testing
- Non-Glenohumeral internal rotation deficit (GIRD) Group: No GIRD (<10° internal rotation deficit)
  Interventions: Other: Glenohumeral Rotation ROM, Shoulder Endurance, and Upper Extremity Stability Testing

INTERVENTIONS:
Other: Glenohumeral Rotation ROM, Shoulder Endurance, and Upper Extremity Stability Testing — Participants undergo a standardized shoulder assessment session. Glenohumeral internal and external rotation range of motion is measured using a goniometric clinical procedure with the shoulder positioned in standardized alignment. Functional performance is assessed using a battery of tests including a shoulder endurance test, a posterior shoulder endurance test, and a modified closed kinetic chain upper extremity stability test. All procedures are performed in a controlled laboratory setting by trained assessors following a consistent protocol.

SUMMARY:
This study aims to investigate whether glenohumeral internal rotation deficit (GIRD) is associated with shoulder endurance and functional stability in male adolescent volleyball players aged 14 to 18 years who do not have shoulder pain. GIRD refers to a reduction in internal rotation range of motion of the dominant (spiking) shoulder compared with the non-dominant shoulder and is commonly observed in young athletes participating in overhead sports such as volleyball.

Participants will be divided into two groups based on shoulder range of motion measurements. Athletes with a loss of at least 10 degrees of internal rotation in the dominant shoulder compared to the non-dominant shoulder will be classified as having GIRD, while those without this difference will be classified as not having GIRD. Shoulder internal and external rotation range of motion will be measured using standardized clinical assessment methods.

Shoulder endurance and upper extremity functional stability will then be evaluated using clinically applicable performance-based tests, including the Shoulder Endurance Test, the Posterior Shoulder Endurance Test, and the Modified Closed Kinetic Chain Upper Extremity Stability Test. The results of these tests will be compared between athletes with and without GIRD.

The main research question of this study is whether the presence of GIRD in asymptomatic adolescent volleyball players is associated with reduced shoulder muscle endurance and decreased functional stability of the upper extremity. The study hypothesizes that athletes with GIRD will demonstrate lower posterior shoulder endurance and poorer upper extremity stability compared to athletes without GIRD.

DETAILED DESCRIPTION:
Repetitive overhead sports activities are known to produce sport-specific adaptations in the glenohumeral joint. One of the most commonly observed adaptations is a reduction in glenohumeral internal rotation on the dominant side, referred to as glenohumeral internal rotation deficit (GIRD). Although GIRD has been widely investigated in adult athletes and in relation to shoulder pain and injury, less is known about its functional implications in asymptomatic adolescent athletes.

This study is designed to explore the association between GIRD and shoulder-related functional performance parameters in adolescent volleyball players. The focus of the protocol is on muscle endurance and dynamic upper extremity stability, which are key components of shoulder function during repetitive overhead tasks. The study specifically examines whether alterations in glenohumeral rotation are reflected in measurable differences in performance-based clinical tests, even in the absence of pain or reported injury.

Standardized physical assessment procedures are used to quantify shoulder rotation and functional performance. All measurements are performed by trained assessors using consistent testing protocols to minimize inter-rater and intra-rater variability. Testing is conducted under controlled laboratory conditions to ensure uniformity across participants.

The analytical approach is based on between-group comparisons according to the presence or absence of GIRD. Statistical methods are selected to evaluate differences in endurance and stability outcomes and to quantify the magnitude of these differences. Sample size estimation is based on previously published data examining shoulder endurance and stability outcomes in overhead athletes.

This protocol aims to contribute to the understanding of early functional changes associated with shoulder motion adaptations in adolescent volleyball players and to inform future injury prevention and training strategies in youth overhead sports.

ELIGIBILITY:
Inclusion Criteria:

* Male adolescent volleyball players aged 14-18 years
* Be a licensed volleyball player for at least 3 years.
* Be male and currently without shoulder symptoms (no current shoulder complaint)

Exclusion Criteria:

* Signs of possible shoulder impingement: 3 or more positive results out of 5 clinical shoulder tests (Neer test, Hawkins-Kennedy test, Painful Arc test 60°-120°, infraspinatus weakness, Empty Can test)
* Shoulder pain within the last 6 months.
* A history of shoulder surgery

Ages: 14 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Eligibility is limited to individuals who are biologically male.
Study Population: The study population consists of adolescent male volleyball players aged 14-18 years with at least 3 years of licensed volleyball experience.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Shoulder Endurance Test (SET) Duration | Through study completion, an average of 1 year
  Shoulder endurance measured as time to volitional fatigue (seconds) during the Shoulder Endurance Test. Participants stand with the back against a wall and perform repeated movements from 90° shoulder flexion to 90° abduction with 90° external rotation and back, using a 1-m green TheraBand anchored to achieve ~100% elongation. Cadence is metronome-controlled and progressively increased (60 bpm, then 90, 120, and 150 bpm). Score range: 0 seconds to no upper limit; higher seconds indicate better endurance.

SECONDARY OUTCOMES:
Posterior Shoulder Endurance Test (PSET) Duration | through study completion, an average of 1 year
  Posterior shoulder endurance measured as time (seconds) the participant can maintain the test position while holding an individually calculated external load. In prone position with the test arm over the table edge, the shoulder is positioned at 90° flexion; the participant elevates the arm to 90° abduction (thumb up) and maintains contact with a level bar apparatus. The test ends if contact is lost or compensatory movements occur. Score range: 0 seconds to no upper limit; higher seconds indicate better posterior shoulder endurance
Modified Closed Kinetic Chain Upper Extremity Stability Test (Modified CKCUEST) Score | through study completion, an average of 1 year
  Upper extremity functional stability measured as the mean number of touches completed in 15 seconds during the Modified Closed Kinetic Chain Upper Extremity Stability Test. Hand placement is standardized using the distance between the acromion processes. From a push-up position, participants alternately touch the dorsal surface of the contralateral hand and return to start as many times as possible. Three trials are performed; the mean of three trials is the score. Score range: 0 touches to no upper limit; higher values indicate better stability.

CONTACTS AND LOCATIONS:
Overall Officials: Seda Bicici Ulusahin, PhD, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Faculty of Physiotherapy and Rehabilitation, University of Health Sciences, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data (IPD) at this time